CLINICAL TRIAL: NCT01465139
Title: A Phase 1 Safety, Pharmacokinetic, and Immunologic Study to Evaluate CDX-301 (rhuFlt3L) in Healthy Volunteers
Brief Title: A Study to Evaluate CDX-301 (rhuFlt3L) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CDX301-02
Record Dates: First submitted 2011-10-13; First posted 2011-11-04 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CDX-301 (Experimental): CDX-301 (rhuFlt3L), administered to healthy patients.
  Interventions: Drug: CDX-301

INTERVENTIONS:
Drug: CDX-301 — CDX-301, administered in multiple dosages and frequencies depending on arm:
  n=3-6 at between 1-75 μg/kg over 5 days
  n=3-6 at 25 μg/kg over 7 days
  n=3-6 at 25 μg/kg over 10 days

SUMMARY:
CDX-301 is a protein that stimulates the growth of bone marrow stem cells and certain immune cells. This study is testing CDX-301 in healthy volunteers who will be monitored for safety and biological response for approximately one month or more.

DETAILED DESCRIPTION:
A total of seven cohorts of healthy volunteers are planned with doses of CDX-301 (rhuFlt3L) ranging between 1 and 75 μg/kg and dosing durations between 5 and 10 days.

Volunteers will be admitted to an inpatient unit during the Treatment Period. Blood samples will be collected periodically to assess the effect of CDX-301. Volunteers will be followed for safety for 28 days following the last dose. Any volunteer who develops anti-CDX-301 antibodies will be followed monthly until the antibody response is below the limit of detection. In general, the total duration of the study will be between approximately 33-38 days.

ELIGIBILITY:
Inclusion Criteria:

Among other criteria, volunteers must meet the following conditions to be eligible for the study:

1. Ages 18 - 55
2. Body Weight ≤ 120 kg
3. Generally good health and without significant medical conditions
4. Willing to use effective method of contraception
5. Abstinence from alcohol for 72 hours prior to study drug administration and throughout the study
6. Negative screening test for HIV, hepatitis B, and hepatitis C
7. Provide written informed consent

Exclusion Criteria:

Among other criteria, volunteers who meet the following conditions are NOT eligible for the study:

1. Drug or alcohol abuse within 12 months
2. Positive drug screen
3. Receipt of certain types of experimental drugs or other treatments, or certain medications
4. Use of systemic immunosuppressive agents (excluding topical steroids) within 12 months
5. History of certain diseases including syphilis, herpes zoster, primary or secondary immunodeficiency
6. Diagnosis with or family history of significant autoimmunity (ex: type I diabetes, multiple sclerosis, rheumatoid arthritis, scleroderma)
7. Any history of cancer, excluding adequately treated and cured basal or squamous cell carcinoma of the skin, or cervical carcinoma in situ within 2 years
8. History of asthma requiring any use of inhaled or oral medication within 5 years
9. Herpes zoster within 3 months
10. Donation of blood within 8 weeks, and donation of plasma within 2 weeks

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number of reported adverse events | Until day 28 of follow up.
  The number of adverse events along with the results of vital sign measurements, physical examinations, and clinical laboratory tests will be used to determine the safety profile of CDX301.

SECONDARY OUTCOMES:
Determination of PK profile of CDX301 | Until day 28 of follow up or until resolution.
  Levels of CDX301 in circulating blood will be evaluated by measures such as AUC, Cmax, T1/2, and Tmax
Immune system effects (eg: anti-CDX-301 antibody development, lymphoid cell populations, serum cytokines, and response to recall antigens and vaccination). | Until day 28 of follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Rockefeller University, New York, New York, United States

REFERENCES:
- [Background] Anandasabapathy N, Breton G, Hurley A, Caskey M, Trumpfheller C, Sarma P, Pring J, Pack M, Buckley N, Matei I, Lyden D, Green J, Hawthorne T, Marsh HC, Yellin M, Davis T, Keler T, Schlesinger SJ. Efficacy and safety of CDX-301, recombinant human Flt3L, at expanding dendritic cells and hematopoietic stem cells in healthy human volunteers. Bone Marrow Transplant. 2015 Jul;50(7):924-30. doi: 10.1038/bmt.2015.74. Epub 2015 Apr 27. PMID 25915810